CLINICAL TRIAL: NCT06974279
Title: Precision Neuromodulation in Post-Stroke Aphasia Using TMS
Brief Title: Post-Stroke Aphasia TMS
Acronym: TaMS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Priyanka Shah-Basak, PhD, Assistant Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRO00053951
Record Dates: First submitted 2025-02-17; First posted 2025-05-15 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Aphasia; Stroke; Language
Keywords: Aphasia; Stroke; Language; TMS
MeSH Terms: conditions — Aphasia; Stroke; Language

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Precision TMS (Active Comparator): SFA will be administered immediately after precision TMS
  Interventions: Device: Precision TMS with SFA
- Control TMS (Placebo Comparator): SFA will be administered immediately after control TMS
  Interventions: Device: Control TMS with SFA

INTERVENTIONS:
Device: Precision TMS with SFA — Excitatory TMS delivered using a precision site finding approach and intermittent theta burst stimulation protocol
  Arms: Precision TMS
Device: Control TMS with SFA — Excitatory TMS using intermittent theta burst stimulation delivered to a control vertex site.
  Arms: Control TMS

SUMMARY:
The investigator proposes to examine the effects of excitatory transcranial magnetic stimulation (TMS) combined with semantic feature analysis (SFA) language therapy to improve word-finding abilities in stroke survivors with aphasia (SWA).

DETAILED DESCRIPTION:
In this project, the investigator will use functional neuroimaging and inhibitory TMS to determine precise therapy-responsive targets for excitatory TMS therapy with SFA. One group of stroke survivors will receive SFA + TMS targeting the precision site, and another group will receive SFA + TMS targeting a control site. The primary outcome will be changes in picture naming accuracy. We expect that excitatory TMS targeting a precision site would result in larger improvements in naming accuracy than TMS targeting a control site. Results will provide the efficacy of precision TMS in post-stroke aphasia.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with left hemisphere stroke
* Consent date >= 1 month after stroke onset
* Fluent in English
* 18 years of age or older

Exclusion Criteria:

* Severe cognitive, auditory or visual impairments that would preclude cognitive and language testing
* Presence of major untreated or unstable psychiatric disease (e.g. schizophrenia, bipolar disease)
* A chronic medical condition that is not treated or is unstable
* The presence of cardiac stimulators or pacemakers or intracardiac lines, neurostimulators, medication infusion device, any other implants near the scalp (e.g., cochlear implants) or in the eye, metal in the body (e.g., splinters, fragments, clips)
* Pregnancy
* History of skull fractures, or skin diseases
* History of ongoing or unmanaged seizures
* Presence of factors that potentially decrease seizure thresholds: on pro-convulsant medications, untreated sleep deprivation or insomnia, ongoing alcoholism or illegal drug abuse (e.g., cocaine or MDMA users)
* History of dyslexia or other developmental learning disabilities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2036-12-31 (Estimated); Study Completion 2036-12-31 (Estimated)

PRIMARY OUTCOMES:
Accuracy on a picture naming test | immediately after and 8-12 weeks after last SFA+TMS treatment
  Changes in accuracy on untrained stimuli after SFA+TMS compared between groups (precision, control).

CONTACTS AND LOCATIONS:
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Patrício, Brígida F, Luis M. T. Jesus and Madeline N. Cruice. "Quality of life of the caregivers of people with aphasia. A systematic review." (2013).
- [Background] Esteban, O., Blair, R., Markiewicz, C. J., Berleant, S. L., Moodie, C., Ma, F., Isik, A. I., Erramuzpe, A., Goncalves, M., Poldrack, R. A., & Gorgolewski, K. J. (2017). poldracklab/fmriprep: 1.0.0-rc5 (1.0.0-rc5). Zenodo. https://doi.org/10.5281/zenodo.996169
- [Background] Hallett M. Transcranial magnetic stimulation: a primer. Neuron. 2007 Jul 19;55(2):187-99. doi: 10.1016/j.neuron.2007.06.026. PMID 17640522
- [Background] Griffis JC, Nenert R, Allendorfer JB, Szaflarski JP. Interhemispheric Plasticity following Intermittent Theta Burst Stimulation in Chronic Poststroke Aphasia. Neural Plast. 2016;2016:4796906. doi: 10.1155/2016/4796906. Epub 2016 Jan 10. PMID 26881111
- [Background] Rossi S, Hallett M, Rossini PM, Pascual-Leone A. Screening questionnaire before TMS: an update. Clin Neurophysiol. 2011 Aug;122(8):1686. doi: 10.1016/j.clinph.2010.12.037. Epub 2011 Jan 11. No abstract available. PMID 21227747
- [Background] Keel JC, Smith MJ, Wassermann EM. A safety screening questionnaire for transcranial magnetic stimulation. Clin Neurophysiol. 2001 Apr;112(4):720. doi: 10.1016/s1388-2457(00)00518-6. No abstract available. PMID 11332408
- [Background] Wassermann EM. Risk and safety of repetitive transcranial magnetic stimulation: report and suggested guidelines from the International Workshop on the Safety of Repetitive Transcranial Magnetic Stimulation, June 5-7, 1996. Electroencephalogr Clin Neurophysiol. 1998 Jan;108(1):1-16. doi: 10.1016/s0168-5597(97)00096-8. PMID 9474057
- [Background] Oberman L, Edwards D, Eldaief M, Pascual-Leone A. Safety of theta burst transcranial magnetic stimulation: a systematic review of the literature. J Clin Neurophysiol. 2011 Feb;28(1):67-74. doi: 10.1097/WNP.0b013e318205135f. PMID 21221011
- [Background] Lerner AJ, Wassermann EM, Tamir DI. Seizures from transcranial magnetic stimulation 2012-2016: Results of a survey of active laboratories and clinics. Clin Neurophysiol. 2019 Aug;130(8):1409-1416. doi: 10.1016/j.clinph.2019.03.016. Epub 2019 Apr 6. PMID 31104898
- [Background] Rossi S, Antal A, Bestmann S, Bikson M, Brewer C, Brockmoller J, Carpenter LL, Cincotta M, Chen R, Daskalakis JD, Di Lazzaro V, Fox MD, George MS, Gilbert D, Kimiskidis VK, Koch G, Ilmoniemi RJ, Lefaucheur JP, Leocani L, Lisanby SH, Miniussi C, Padberg F, Pascual-Leone A, Paulus W, Peterchev AV, Quartarone A, Rotenberg A, Rothwell J, Rossini PM, Santarnecchi E, Shafi MM, Siebner HR, Ugawa Y, Wassermann EM, Zangen A, Ziemann U, Hallett M; basis of this article began with a Consensus Statement from the IFCN Workshop on "Present, Future of TMS: Safety, Ethical Guidelines", Siena, October 17-20, 2018, updating through April 2020. Safety and recommendations for TMS use in healthy subjects and patient populations, with updates on training, ethical and regulatory issues: Expert Guidelines. Clin Neurophysiol. 2021 Jan;132(1):269-306. doi: 10.1016/j.clinph.2020.10.003. Epub 2020 Oct 24. PMID 33243615
- [Background] Rossi S, Hallett M, Rossini PM, Pascual-Leone A; Safety of TMS Consensus Group. Safety, ethical considerations, and application guidelines for the use of transcranial magnetic stimulation in clinical practice and research. Clin Neurophysiol. 2009 Dec;120(12):2008-2039. doi: 10.1016/j.clinph.2009.08.016. Epub 2009 Oct 14. PMID 19833552
- [Background] Radford, A., Kim, J. W., Xu, T., Brockman, G., McLeavey, C., & Sutskever, I. (2023). Robust speech recognition via large-scale weak supervision. Proceedings of the 40th International Conference on Machine Learning, 202, 28492-28518.
- [Background] Wilson SM, Eriksson DK, Schneck SM, Lucanie JM. A quick aphasia battery for efficient, reliable, and multidimensional assessment of language function. PLoS One. 2018 Feb 9;13(2):e0192773. doi: 10.1371/journal.pone.0192773. eCollection 2018. PMID 29425241
- [Background] Lin Y, Zhu M, Su Z. The pursuit of balance: An overview of covariate-adaptive randomization techniques in clinical trials. Contemp Clin Trials. 2015 Nov;45(Pt A):21-5. doi: 10.1016/j.cct.2015.07.011. Epub 2015 Aug 2. PMID 26244705
- [Background] Walsh V, Cowey A. Transcranial magnetic stimulation and cognitive neuroscience. Nat Rev Neurosci. 2000 Oct;1(1):73-9. doi: 10.1038/35036239. PMID 11252771
- [Background] Devlin JT, Watkins KE. Stimulating language: insights from TMS. Brain. 2007 Mar;130(Pt 3):610-22. doi: 10.1093/brain/awl331. Epub 2006 Nov 29. PMID 17138570
- [Background] Pascual-Leone A, Bartres-Faz D, Keenan JP. Transcranial magnetic stimulation: studying the brain-behaviour relationship by induction of 'virtual lesions'. Philos Trans R Soc Lond B Biol Sci. 1999 Jul 29;354(1387):1229-38. doi: 10.1098/rstb.1999.0476. PMID 10466148
- [Background] Vines BW, Schnider NM, Schlaug G. Testing for causality with transcranial direct current stimulation: pitch memory and the left supramarginal gyrus. Neuroreport. 2006 Jul 17;17(10):1047-50. doi: 10.1097/01.wnr.0000223396.05070.a2. PMID 16791101
- [Background] Fridriksson J, Rorden C, Elm J, Sen S, George MS, Bonilha L. Transcranial Direct Current Stimulation vs Sham Stimulation to Treat Aphasia After Stroke: A Randomized Clinical Trial. JAMA Neurol. 2018 Dec 1;75(12):1470-1476. doi: 10.1001/jamaneurol.2018.2287. PMID 30128538
- [Background] Abo M, Kakuda W, Watanabe M, Morooka A, Kawakami K, Senoo A. Effectiveness of low-frequency rTMS and intensive speech therapy in poststroke patients with aphasia: a pilot study based on evaluation by fMRI in relation to type of aphasia. Eur Neurol. 2012;68(4):199-208. doi: 10.1159/000338773. Epub 2012 Aug 29. PMID 22948550
- [Background] Lefaucheur JP, Aleman A, Baeken C, Benninger DH, Brunelin J, Di Lazzaro V, Filipovic SR, Grefkes C, Hasan A, Hummel FC, Jaaskelainen SK, Langguth B, Leocani L, Londero A, Nardone R, Nguyen JP, Nyffeler T, Oliveira-Maia AJ, Oliviero A, Padberg F, Palm U, Paulus W, Poulet E, Quartarone A, Rachid F, Rektorova I, Rossi S, Sahlsten H, Schecklmann M, Szekely D, Ziemann U. Evidence-based guidelines on the therapeutic use of repetitive transcranial magnetic stimulation (rTMS): An update (2014-2018). Clin Neurophysiol. 2020 Feb;131(2):474-528. doi: 10.1016/j.clinph.2019.11.002. Epub 2020 Jan 1. PMID 31901449
- [Background] Hamilton RH, Chrysikou EG, Coslett B. Mechanisms of aphasia recovery after stroke and the role of noninvasive brain stimulation. Brain Lang. 2011 Jul;118(1-2):40-50. doi: 10.1016/j.bandl.2011.02.005. Epub 2011 Apr 2. PMID 21459427
- [Background] Shah-Basak PP, Wurzman R, Purcell JB, Gervits F, Hamilton R. Fields or flows? A comparative metaanalysis of transcranial magnetic and direct current stimulation to treat post-stroke aphasia. Restor Neurol Neurosci. 2016 May 2;34(4):537-58. doi: 10.3233/RNN-150616. PMID 27163249
- [Background] Norise C, Hamilton RH. Non-invasive Brain Stimulation in the Treatment of Post-stroke and Neurodegenerative Aphasia: Parallels, Differences, and Lessons Learned. Front Hum Neurosci. 2017 Jan 23;10:675. doi: 10.3389/fnhum.2016.00675. eCollection 2016. PMID 28167904
- [Background] Kielar A, Patterson D, Chou YH. Efficacy of repetitive transcranial magnetic stimulation in treating stroke aphasia: Systematic review and meta-analysis. Clin Neurophysiol. 2022 Aug;140:196-227. doi: 10.1016/j.clinph.2022.04.017. Epub 2022 May 5. PMID 35606322
- [Background] Chou TY, Wang JC, Lin MY, Tsai PY. Low-Frequency vs. Theta Burst Transcranial Magnetic Stimulation for the Treatment of Chronic Non-fluent Aphasia in Stroke: A Proof-of-Concept Study. Front Aging Neurosci. 2022 Jan 14;13:800377. doi: 10.3389/fnagi.2021.800377. eCollection 2021. PMID 35095477
- [Background] Huang YZ, Edwards MJ, Rounis E, Bhatia KP, Rothwell JC. Theta burst stimulation of the human motor cortex. Neuron. 2005 Jan 20;45(2):201-6. doi: 10.1016/j.neuron.2004.12.033. PMID 15664172
- [Background] Chen R, Classen J, Gerloff C, Celnik P, Wassermann EM, Hallett M, Cohen LG. Depression of motor cortex excitability by low-frequency transcranial magnetic stimulation. Neurology. 1997 May;48(5):1398-403. doi: 10.1212/wnl.48.5.1398. PMID 9153480
- [Background] Shah-Basak PP, Norise C, Garcia G, Torres J, Faseyitan O, Hamilton RH. Individualized treatment with transcranial direct current stimulation in patients with chronic non-fluent aphasia due to stroke. Front Hum Neurosci. 2015 Apr 21;9:201. doi: 10.3389/fnhum.2015.00201. eCollection 2015. PMID 25954178
- [Background] Paulus W. Toward establishing a therapeutic window for rTMS by theta burst stimulation. Neuron. 2005 Jan 20;45(2):181-3. doi: 10.1016/j.neuron.2005.01.008. PMID 15664167
- [Background] Szaflarski JP, Nenert R, Allendorfer JB, Martin AN, Amara AW, Griffis JC, Dietz A, Mark VW, Sung VW, Walker HC, Zhou X, Lindsell CJ. Intermittent Theta Burst Stimulation (iTBS) for Treatment of Chronic Post-Stroke Aphasia: Results of a Pilot Randomized, Double-Blind, Sham-Controlled Trial. Med Sci Monit. 2021 Jun 29;27:e931468. doi: 10.12659/MSM.931468. PMID 34183640
- [Background] Szaflarski JP, Griffis J, Vannest J, Allendorfer JB, Nenert R, Amara AW, Sung V, Walker HC, Martin AN, Mark VW, Zhou X. A feasibility study of combined intermittent theta burst stimulation and modified constraint-induced aphasia therapy in chronic post-stroke aphasia. Restor Neurol Neurosci. 2018;36(4):503-518. doi: 10.3233/RNN-180812. PMID 29889086
- [Background] Szaflarski JP, Vannest J, Wu SW, DiFrancesco MW, Banks C, Gilbert DL. Excitatory repetitive transcranial magnetic stimulation induces improvements in chronic post-stroke aphasia. Med Sci Monit. 2011 Feb 25;17(3):CR132-9. doi: 10.12659/msm.881446. PMID 21358599
- [Background] Shah-Basak P, Boukrina O, Li XR, Jebahi F, Kielar A. Targeted neurorehabilitation strategies in post-stroke aphasia. Restor Neurol Neurosci. 2023;41(3-4):129-191. doi: 10.3233/RNN-231344. PMID 37980575